# What are the Patterns of Patient Engagement Trends in Stave IV Melanoma Clinical Trials?

This is an Informed Consent Form For Stave IV Melanoma Patients in <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: October 15, 2023

Understanding the Importance of This Consent Form

If you are in the process of filling out this paperwork, it suggests that you might qualify to take part in a distinctive observational clinical study designed specifically for individuals with stage IV melanoma. This detailed handbook elucidates the primary objectives of the study, the intricate execution strategy, and the various implications, encompassing both favorable and potentially unfavorable consequences. Before reaching a decision, it is crucial to thoroughly examine the specifics of your potential involvement, and seeking guidance from a reliable source can offer invaluable insights. If any segment of this document seems perplexing or if you have inquiries, rest assured that the researcher is accessible to provide explanations.

Understanding the Significance of Stage IV Melanoma Clinical Trials

Stage IV melanoma is the most advanced stage of melanoma, a type of skin cancer. At this stage, the cancer has spread from the skin to distant parts of the body, such as distant lymph nodes, the lungs, liver, brain, or other organs. Stage IV melanoma is considered to be metastatic and is more challenging to treat than earlier stages. Treatment options for stage IV melanoma may include surgery, immunotherapy, targeted therapy, chemotherapy, or radiation therapy, depending on the location and extent of the metastases

Clinical trials, specifically focused on stage IV melanoma, are crucial in assessing the safety and efficacy of new treatments for this disease. These trials serve as fundamental instruments in determining whether emerging medications outperform standard therapies, providing compelling evidence to support their wider implementation.

What distinguishes this particular study is its primary emphasis on the real-life experiences of individuals grappling with stage IV melanoma, actively engaging in a clinical trial involving medical interventions. The main goal is to thoroughly scrutinize trial completion rates and voluntary withdrawals among this particular group of patients.

#### Delving into the Essence of Observational Clinical Trials

Engaging in this medical trial involves immersing yourself in an observational study, a distinct feature of clinical research meticulously crafted to gather insights through unobtrusive observation of patients while preserving their treatment plans.

Researchers will solely observe your journey, meticulously assessing the outcomes of your condition without making any alterations. This trial design is crucial in enhancing our understanding of the intrinsic progression of a specific medical ailment and its implications for those affected by it. Your active participation in this observational study is integral to expanding the boundaries of medical knowledge and propelling advancements in the care provided to individuals with the same condition.

# Distinguishing This Study from Other Stage IV Melanoma Clinical Trials

Understanding the unique aspects of this research investigation is crucial. It operates solely on an observational basis, implying that your participation will not involve any specific treatments or interventions. To arrive at an informed decision about potential participation in a clinical trial, it is essential to comprehend the spectrum of stage IV melanoma clinical research, including interventional studies where participants undergo various treatment regimens.

Crafting an informed decision about your potential involvement in a clinical trial requires an active approach that entails research and comparison of trials. Platforms such as Clinicaltrials.gov and similar sites provide a wealth of information on <a href="stage-IV melanoma">stage-IV melanoma</a> research. Additionally, Power's specialized online platform offers a comprehensive list of ongoing <a href="stage-IV melanoma clinical trials">stage-IV melanoma clinical trials</a> actively recruiting volunteers. Equipped with

thorough research and a comprehensive understanding of different clinical trial categories, you can confidently shape your participation decision.

## Safeguarding the Privacy of Your Data

Throughout this research initiative, the safeguarding of your data's complete confidentiality remains a top priority. To ensure your anonymity, we kindly urge you to refrain from providing any personal or identifiable information in your responses to the questionnaires. The research team is resolute in its efforts to strengthen the security of your privacy. Nevertheless, it is important to note that specific legal situations may arise, requiring the release of personal data.

### **Engaging in Clinical Trial Surveys**

You are invited to actively participate in this observational clinical study by sharing your experiences. Your involvement will entail the completion of surveys every two weeks, taking up approximately 20-30 minutes of your time. Additionally, we have established regular check-in calls every quarter, ensuring ongoing support and communication throughout your participation.

It is essential to highlight the voluntary nature of your participation in the survey phase of the trial. You have the freedom to respond to specific questions or complete the entire questionnaire as you see fit. Moreover, you retain the right to withdraw from the trial at any point. Recognizing the personal significance of enrolling in a clinical trial, we are dedicated to providing the necessary guidance, valuing your privacy, and supporting your decision-making process throughout the trial.

## Anticipated Advantages in Perspective

Although immediate benefits may not be readily apparent to those engaged in this observational clinical research, their involvement holds the potential to significantly influence others. The data collected from participants will serve to improve future approaches to engaging individuals with stage IV melanoma, potentially expanding the horizons of medical research. Those who embark on this journey of treatment have the capacity to instigate transformative changes in medical research, possibly shaping the future for those grappling with stage IV melanoma.

#### Acknowledging Potential Health Implications

Despite the significant strides made in clinical trials, it remains essential to acknowledge the potential health implications that participants might encounter, particularly in trials evaluating new medications.

Nevertheless, our methodology in observational clinical research adopts a distinct approach, mitigating these risks by abstaining from the administration of experimental drugs to participants. Instead, our primary emphasis lies in comprehensive monitoring and evaluating outcomes, ensuring the prevention of any unwarranted health hazards.

#### Promoting Diversity in Clinical Research

A wealth of online resources eagerly anticipates your active engagement if you possess an unyielding curiosity to explore the multifaceted realm of diversity in clinical trials.

Whether your aim is to comprehend the intricacies of the challenges and opportunities associated with clinical trial diversity or to expand your personal perspectives, the following resources can prove invaluable:

Ramos, Edward, Katie Baca-Motes, Jay A. Pandit, and Toluwalase A. Ajayi. "Improving participant representation in the era of digital clinical studies." *Trends in Molecular Medicine* (2022).

Hurwitz, Brian. "Form and representation in clinical case reports." *Literature and Medicine* 25, no. 2 (2006): 216-240.

# Confirmation of Informed Participation

I hereby affirm that I have dedicated ample time to comprehending and absorbing the information provided in the informed consent form. This understanding has been achieved through either independent review or guidance from a trusted individual who has elucidated its contents to me. All of my concerns and queries have been thoroughly addressed to my utmost satisfaction.

I am well aware that my involvement in this study is entirely of my own volition, and I retain the sole right to revoke my consent without the need to provide explanations or bear any financial obligations. It has been made clear to me that I will be provided with a copy of this informed consent form for my personal records.

After careful consideration and thorough examination of all the material presented to me, I hereby extend my consent to participate in this study, reflecting my informed and independent decision.

| Participant Name |
|-----------------------|
| · |
| Participant Signature |
| Date |

## Affirmation by Informed Consent Facilitator

I affirm that I conducted an exhaustive discussion with the participant, meticulously elucidating the intricacies outlined in this written document. My objective was to ensure that the participants comprehensively understood the primary study objectives, methodologies employed, potential risks and benefits, and other critical aspects of the stage IV melanoma clinical trial.

The participant was afforded sufficient opportunity to raise questions, express concerns, and seek clarification. It is imperative to emphasize that the participant's involvement in this study is entirely voluntary, and they retain the unrestricted right to withdraw at any time, for any reason, without assuming any financial responsibilities.

Following the participant's consent, a meticulously preserved copy of this written document was provided, serving as a repository for their personal information.

| Printed Name of Assisting Researcher |
|--------------------------------------|
| Signature of Assisting Researcher |
| Date |